CLINICAL TRIAL: NCT02262364
Title: A Pilot Study of a Single Intra-articular Injection of Autologous Protein Solution in Patients With Knee Osteoarthritis
Brief Title: Safety of NStride Autologous Protein Solution in the Treatment of Knee Osteoarthritis (PROGRESS I)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Collaborators: Biomet Biologics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APSS-22-01
Record Dates: First submitted 2014-09-19; First posted 2014-10-13 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2018-10

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NStride APS (Experimental): Subjects will receive an intra-articular injection of APS.
  Interventions: Biological: APS

INTERVENTIONS:
Biological: APS — See above

SUMMARY:
The primary objective of this study is to assess the safety of a single injection of APS.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the safety of a single injection of APS in patients with painful unilateral knee osteoarthritis and who have not been able to get satisfactory pain relief with other treatments through one-month post treatment and monitor subjects for adverse events through 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥40 and ≤75 years old at time of injection..
* A standing radiograph of the knee showing a Kellgren-Lawrence grade of 2 to 4 (within 6 months of screening).
* Body mass index ≤40 kg/m2.
* A Western Ontario and McMaster Universities osteoarthritis index using the Likert scale, Version 3. (WOMAC LK 3.1) pain subscale total score ≥ 10 and ≤ 19.
* Has undergone at least two prior conservative OA therapies without satisfactory pain relief.
* Patient has failed to get satisfactory pain relief from either HA or steroid injections or would be considered an appropriate patient to receive either HA or steroid injections

Exclusion Criteria:

* Presence of active infection or abnormal effusion in the knee immediately preceding treatment injection.
* Presence of symptomatic OA in the non-study knee
* Diagnosed with rheumatoid arthritis, Reiter's syndrome, psoriatic arthritis, gout, ankylosing spondylitis, chondromalacia, arthritis secondary to other inflammatory diseases, or of metabolic origin; HIV, viral hepatitis; chondrocalcinosis, Paget's disease, villonodular synovitis, and other non-OA joint disease.
* Disease of spine, hip or other lower extremity joints of sufficient degree to affect assessment of the index knee
* Untreated symptomatic injury of index knee (e.g., acute traumatic injury, anterior cruciate ligament injury, meniscus injury, cartilage lesion).
* Knee radiographs showing bone-on-bone or other gross cartilage deficits.
* Presence of surgical hardware or other foreign body in the index knee.
* Intra-articular steroid injections in the index knee within 3 months of screening.
* Intra-articular HA in the index knee within 6 months of screening.
* Other intra-articular therapy in the index knee within 6 months prior to screening.
* Systemic steroid use within 2 weeks of screening.
* Planned/anticipated surgery of the index knee during the study period.
* A history of local anesthetic allergy
* Use of systemic immunosuppressants within six weeks of treatment.
* Currently on anticoagulant therapy
* Any documented clinically significant condition (e.g., diabetes, malignancy), finding, or psychiatric illness at screening which could compromise patient safety or interfere with the assessment of the safety and treatment effects of the study injection.
* Skin breakdown at the index knee where the injection is planned to take place.
* Pregnant or nursing mothers or women who are planning on getting pregnant during the time they will be participating in the study.
* Known drug or alcohol dependence currently or within the last year.
* Used any investigational drug or device within 30 days prior to screening.
* Used any investigational biologic within 60 days prior to screening

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Klaassen, Principal Investigator — OSMC
Locations (1):
- Orthopedic and Sports Medicine Center of Northern Indiana (OSMC), Elkhart, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Period: Study Enrollment
Arm/Group | NStride APS
Started | 11
Completed | 11
Not Completed | 0
Period: Blood Draw for Device Processing
Arm/Group | NStride APS
Started | 11
Completed | 10
Not Completed | 1
Not completed — Insufficient blood could be drawn | 1
Period: Injection With APS
Arm/Group | NStride APS
Started | 10
Completed | 10
Not Completed | 0
Period: Follow-Up Through 12 Months
Arm/Group | NStride APS
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The included population could generally be characterized as patients with painful unilateral knee OA, who had not been able to get satisfactory pain relief with other treatments.
Arm/Group | NStride APS
Number analyzed (Participants) | 10
Age, Customized [Mean (Standard Deviation); unit: years]
  Mean Patient Age | 58.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Description: Adverse Events and Serious Adverse Events
Time Frame: 1 Year
Measure: Number; unit: events
Arm/Group | NStride APS
Number analyzed (Participants) | 10
events
  Adverse Events | 27
  Serious Adverse Events | 1

2. Secondary Outcome: Change From Baseline to 12 Months in Pain, Stiffness, and Function in Daily Living Measured With WOMAC Questionnaire
Description: The WOMAC LK 3.1 questionnaire is a validated tool commonly used for assessing knee pain, stiffness, and function. The WOMAC LK 3.1 questionnaire has 24 items that the patient addresses about the knee: 5 items on the pain subscale, 2 on the stiffness subscale, and 17 on the physical function subscale. Each item is answered on a 5-point Likert scale, with grading from 0 (none or never) to 4 (extreme or always). A higher score indicates worse pain, stiffness, or functional limitation.
  The WOMAC pain subscale consists of five questions scored from 0 to 4. The pain score has a range of 0 (no pain) to 20 (maximal pain).
  The WOMAC stiffness subscale consists of two questions scored from 0 to 4. The stiffness score has a range of 0 (no stiffness) to 8 (maximal stiffness).
  The WOMAC physical function subscale consists of seventeen questions scored from 0 to 4. The physical function score has a range of 0 (no functional limitation) to 68 (maximal functional limitation).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NStride APS
Number analyzed (Participants) | 10
units on a scale
  WOMAC Pain - Baseline | 12.2 (1.7)
  WOMAC Pain - 12 Months | 3.3 (2.9)
  WOMAC Stiffness - Baseline | 4.8 (1.4)
  WOMAC Stiffness - 12 Months | 1.6 (1.7)
  WOMAC Physical Function - Baseline | 38.6 (9.4)
  WOMAC Physical Function - 12 Months | 12.1 (9.8)

3. Secondary Outcome: Change From Baseline to 12 Months in Pain as Measured by the Numeric Rating Scale (NRS)
Description: The Numeric Rating Scale (NRS) is a validated measure of knee pain. The NRS is an 11 point Likert type scale anchored by 0 "no pain" and 10 "worst possible pain". Subjects rate their average pain over the last 24 hours.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NStride APS
Number analyzed (Participants) | 10
units on a scale
  NRS Pain - Baseline | 5.9 (1.9)
  NRS Pain - 12 Months | 1.6 (1.6)

4. Secondary Outcome: Change From Baseline to 12 Months in Pain as Measured With Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: The KOOS questionnaire is a commonly used instrument to assess the patient's opinion about their knee and associated problems. KOOS consists of 5 subscales: Pain (9 questions), Symptoms (7 questions), Function in daily living (ADL) (17 questions), Function in sport and recreation (Sport/Rec) (5 questions) and knee related Quality of Life (QOL) (4 questions). The previous week is used as the time period for answering the questions.
  A higher score on the KOOS questionnaire indicates fewer problems, and 0 indicates extreme problems. Each subscale score is calculated independently. The mean score of the individual items of each subscale is calculated and divided by 4 (the highest possible score for a single answer option). Traditionally in orthopedics, 100 indicates no problems and 0 indicates extreme problems. The normalized score is transformed to meet this standard.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NStride APS
Number analyzed (Participants) | 10
units on a scale
  KOOS Pain - Baseline | 36.9 (16.2)
  KOOS Pain - 1 Week | 56.7 (16.5)
  KOOS Pain - 12 Months | 79.7 (16.2)

ADVERSE EVENTS:
Arm/Group | NStride APS
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 7/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NStride APS (N=10)
Diverticulitis (Gastrointestinal disorders) | 1 — The event was considered not related to the device and not related to the procedure
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NStride APS (N=10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Hypertension (Cardiac disorders) | 1
Gingival swelling (General disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Blood glucose increased (Endocrine disorders) | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1
Foot fracture (Musculoskeletal and connective tissue disorders) | 1
Nasopharyngitis (General disorders) | 1
Tooth extraction (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator must provide the Sponsor at least 90 days to review publications for legal and regulatory compliance and will include in publications a statement that the study was supported by the Sponsor. Sponsor confidential information will not be submitted for publication without Sponsor consent. Sponsor may request delay of publication for 60 days to allow for patent application filing.